CLINICAL TRIAL: NCT00598156
Title: Avastin and Chemotherapy Followed by Avastin Alone or in Combination With Tarceva for the Treatment of Metastatic Colorectal Cancer.
Brief Title: Chemotherapy and Avastin Followed by Maintenance Treatment With Avastin +/- Tarceva
Acronym: ACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19033; EUDRACT 2006-002295-18
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Erlotinib Hydrochloride; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): bevacizumab and chemotherapy (according to investigators choice) during 18 weeks, followed by bevacizumab and erlotinib as maintenance treatment until progression
  Interventions: Drug: erlotinib (Tarceva); Drug: bevacizumab (Avastin)
- 2 (Experimental): bevacizumab and chemotherapy (according to investigators choice) during 18 weeks, followed by bevacizumab every third week until progression
  Interventions: Drug: bevacizumab (Avastin)

INTERVENTIONS:
Drug: erlotinib (Tarceva) — Chemotherapy for 18 weeks (XELOX, XELIRI, FOLFOX or FOLFIRI)
  Arms: 1
Drug: bevacizumab (Avastin) — Chemotherapy for 18 weeks (XELOX, XELIRI, FOLFOX or FOLFIRI)

SUMMARY:
Chemotherapy and bevacizumab is given for 4 months. Patients who have not progressed will continue with maintenance treatment with either bevacizumab (Avastin) alone, or bevacizumab and erlotinib (Tarceva).

DETAILED DESCRIPTION:
Patients with metastatic colorectal cancer will be treated with standard chemotherapy according to the investigators choice. In addition to chemotherapy, Avastin (bevacizumab) will be given during the treatment period. After the chemotherapy is finished (after 18 weeks), maintenance therapy will be given and the patients will be randomized to treatment with either with Avastin alone or Avastin in combination with Tarceva (erlotinib). Patients with progressive disease, or patients suitable to curative resection of metastases will be taken out of study.

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma of the colon or rectum.
2. Age > 18.
3. Measurable disease according to RECIST criteria.
4. Expected survival more than three months.
5. Adequate bone marrow, liver and kidney function.
6. INR < 1.5 times upper limit.
7. Adequate contraception for fertile patients.
8. Signed written informed consent.

Exclusion Criteria:

1. Earlier chemotherapy for metastatic colorectal cancer.
2. Adjuvant treatment within 6 months.
3. Surgery or significant trauma within 28 days prior to study entry.
4. Planned radiotherapy against target lesions.
5. CNS metastases.
6. Prior malignancy within 5 years except ca in situ of cervix and basal cell carcinoma.
7. Bleeding diathesis
8. Uncontrolled hypertension.
9. Significant cardiovascular disease.
10. Treatment with anticoagulant drugs.
11. Participation in other clinical trial.
12. Pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2007-06; Primary Completion 2009-10 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 3 years

SECONDARY OUTCOMES:
overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anders Johnsson, MD PhD, Principal Investigator — Lund University Hospital, Sweden
Locations (15):
- Denmark (6):
  - Vejle Hospital, Department of Oncology, Copenhagen
  - Esbjerg Hospital, Esbjerg
  - Herning Hospital, Herning
  - Hillerod Hospital, Department of Oncology, Hillerød
  - Odense Hospital, Department of Oncology, Odense
  - Roskilde Hospital, Department of Oncology, Roskilde
- Sweden (9):
  - Ryhov Hospital, Department of Oncology, Jönköping
  - Kalmar Hospital, Department of Oncology, Kalmar
  - Lund University Hospital, Department of Oncology, Lund
  - University Hospital MAS, Malmo
  - Karolinska University Hospital, Department of Oncology, Stockholm
  - Sundsvall Hospital, Department of Oncology, Sundsvall
  - University Hospital of Norrland, Department of Oncology, Umeå
  - Akademiska Hospital, Department of Oncology, Uppsala
  - Vaxjo Hospital, Department of Oncology, Vaxjo

REFERENCES:
- [Derived] Hansen TF, Christensen Rd, Andersen RF, Sorensen FB, Johnsson A, Jakobsen A. MicroRNA-126 and epidermal growth factor-like domain 7-an angiogenic couple of importance in metastatic colorectal cancer. Results from the Nordic ACT trial. Br J Cancer. 2013 Sep 3;109(5):1243-51. doi: 10.1038/bjc.2013.448. Epub 2013 Aug 6. PMID 23922111
- [Derived] Johnsson A, Hagman H, Frodin JE, Berglund A, Keldsen N, Fernebro E, Sundberg J, De Pont Christensen R, Garm Spindler KL, Bergstrom D, Jakobsen A. A randomized phase III trial on maintenance treatment with bevacizumab alone or in combination with erlotinib after chemotherapy and bevacizumab in metastatic colorectal cancer: the Nordic ACT Trial. Ann Oncol. 2013 Sep;24(9):2335-41. doi: 10.1093/annonc/mdt236. Epub 2013 Jun 19. PMID 23788755